CLINICAL TRIAL: NCT02862691
Title: A Comparison of the Analgesic Efficacy of Oral Opioid Medication vs. Injected Local Anesthetic in Emergency Department Patients With Toothache
Brief Title: Percocet vs. Bupivicaine for Toothaches in the ED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, Vice Chairman of Reserach, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 901314-2
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Toothache
Keywords: toothache
MeSH Terms: conditions — Toothache | interventions — Acetaminophen; Oxycodone; Analgesics; oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral analgesic (Active Comparator): 2 tablets of acetaminophen 325 mg/ oxycodone 5 mg orally once
  Interventions: Drug: Acetaminophen/Oxycodone (Oral analgesic)
- Injectable local anesthetic (Experimental): local injection or nerve block with bupivicaine 0.5%
  Interventions: Drug: Bupivicaine (Injectable local anesthetic)

INTERVENTIONS:
Drug: Acetaminophen/Oxycodone (Oral analgesic) — 2 oral tablets of acetaminophen 325 mg plus oxycodone 5 mg given once
  Other Names: Acetaminophen/Oxycodone
  Arms: Oral analgesic
Drug: Bupivicaine (Injectable local anesthetic) — local injection of bupivicaine 0.5% at root of maxillary tooth or nerve block for mandibular tooth
  Other Names: Bupivicaine
  Arms: Injectable local anesthetic

SUMMARY:
The goal of this study is to compare the speed and adequacy of pain relief in Emergency Department patients with a toothache after an oral analgesic or a local anesthetic administered as a nerve block or by local infiltration.

DETAILED DESCRIPTION:
All adult patients reporting to the Stony Brook Medical Center Emergency Department with a toothache will be assessed for inclusion criteria. Patients who agree to participate in the study and meet the study criteria will be asked to rate their pain using an 11-item verbal numeric pain scale from 0 to 10, from none to worst. The patient will then be randomized to either two Percocet oral tablets (acetaminophen 325 mg and oxycodone 5 mg), or a single dose of Bupivicaine (as a root block for maxillary teeth or as a local infiltration for mandibular teeth). The intervention given to any particular patient will be determined using a randomization protocol described in Treatment Allocation. The patients will be stratified into depending on whether they have mandibular or maxillary tooth pain in order to account for any difference in outcome based on method of Bupivicaine administration (local block for maxillary teeth and nerve block for mandibular teeth). Half of the included patients will have maxillary toothaches and half will have mandibular toothaches. Administration of additional prescriptions and recommendations will be given as deemed necessary by the dental resident and attending physician (such as antibiotics or additional analgesics).

Measures and Outcomes Following the administration of treatment, the patient will be asked to rate their pain on the verbal numeric pain scale every 5 minutes up to 30 minutes following treatment. The pain of injection will also be measured, immediately following injection on the same pain scale. If after the first 30 minutes the patient still requires additional analgesia, then other analgesic interventions may be given at the discretion of the dental resident and attending physician.

The primary outcome will be the percentage of patients with significant pain relief at the end of the study period of 30 minutes. Patients whose pain is reduced from severe (7-10) to mild (0-3) will be considered as having a meaningful reduction in pain. Secondary outcomes will be the absolute change in pain severity at 30 minutes calculated by subtracting the 30-minute pain score from the initial pre-treatment pain score as well as the time to a 50% reduction in pain severity.

At the end of the trial patient satisfaction with the method of analgesia will be measured on a 5 point Likert scale: extremely dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, and extremely satisfied. Patients will also be asked if they would choose the same treatment for future toothaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the ED with a chief complaint of toothache, and a pain intensity rating of at least a 7 on an 11 item verbal numeric scale (from 0 or no pain to 10 or worst imaginable pain) will be eligible for enrollment.
* Patient should have the capacity to provide informed consent.

Exclusion Criteria:

* Patients presenting with a toothache due to trauma or post-operative procedure will be excluded as well as those requiring drainage of a dental abscess.
* Patients who have any contraindications to the medications used in the study (allergy, history of GI bleeding, etc.).
* Patients who cannot remain in the ED for at least 1 hour after study drug administration or do not have a ride home (if receiving Percocet) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with significant pain relief at the end of the study period | 60 minutes
  Patients whose pain is reduced from severe (7-10) to mild (0-3) will be considered as having a meaningful reduction in pain.

SECONDARY OUTCOMES:
Absolute change in pain severity | 60 minutes
  Calculated by subtracting the 60-minute pain score from the initial pre-treatment pain score
The time to a 50% reduction in pain severity | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Singer, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes